CLINICAL TRIAL: NCT00084864
Title: A Pilot Trial of Calcitriol in Localized Prostate Cancer: Investigation of Biologic Effects and Potential Intermediate Endpoints
Brief Title: Calcitriol and Dexamethasone Before Radical Prostatectomy in Treating Patients With Localized Adenocarcinoma (Cancer) of the Prostate
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sample size is too small to draw a conclusion
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP 02-12; P30CA016056 (NIH); RPCI-RP-0212
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Calcitriol; Dexamethasone; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Stage 1, Arm I (Experimental): Patients receive oral dexamethasone once daily on days 1-4 and oral calcitriol once daily on days 2-4 weekly for 4 weeks before surgery.
  Interventions: Dietary Supplement: calcitriol; Drug: dexamethasone
- Stage 1, Arm II (Experimental): No study drugs before surgery.
  Interventions: Other: clinical observation
- Stage 1 Arm 3 (Experimental): Patients receive oral dexamethasone once daily on days 1-4.
  Interventions: Drug: dexamethasone
- Stage 1, Arm 4 (Experimental): Patients receive oral calcitriol once daily on days 2-4.
  Interventions: Dietary Supplement: calcitriol

INTERVENTIONS:
Dietary Supplement: calcitriol — Given orally
  Arms: Stage 1, Arm 4; Stage 1, Arm I
Drug: dexamethasone — Given orally
  Arms: Stage 1 Arm 3; Stage 1, Arm I
Other: clinical observation — No intervention before surgery
  Arms: Stage 1, Arm II

SUMMARY:
RATIONALE: Calcitriol and dexamethasone may slow the growth of prostate cancer cells.

PURPOSE: This randomized phase II trial is studying how well giving calcitriol together with dexamethasone before radical prostatectomy works in treating patients with localized stage II or stage III adenocarcinoma (cancer) of the prostate.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of calcitriol and dexamethasone before radical prostatectomy on tumor vessel density in patients with localized adenocarcinoma of the prostate.
* Determine the effect of this regimen on the extent of prostatic intraepithelial neoplasia in these patients.
* Determine the effect of this regimen on the expression of apoptosis markers, p21, p27, prostate-specific antigen (PSA), prostate-specific membrane antigen, and VDR expression in tumor-associated vascular endothelial cells and endothelium derived from normal-appearing prostate and tumor in these patients.
* Determine the acute effects of this regimen on serum PSA in these patients.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a two-stage, randomized, pilot study.

* Stage 1: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral dexamethasone once daily on days 1-4 and oral calcitriol once daily on days 2-4 weekly for 4 weeks before surgery. Within 48 hours of the last dose, patients undergo radical prostatectomy.
  * Arm II: Patients receive no study drugs, but undergo radical prostatectomy.
* Stage 2: If sufficient activity is seen with the dexamethasone and calcitriol regimen in stage 1, the study is expanded and additional patients are randomized to 1 of 4 treatment arms.

  * Arm I: Patients receive dexamethasone and calcitriol as in stage 1, arm I.
  * Arm II: Patients receive oral dexamethasone once daily on days 1-4.
  * Arm III: Patients receive oral calcitriol once daily on days 2-4.
  * Arm IV: Patients undergo radical prostatectomy as in stage 1, arm II. In arms I, II, and III, patients undergo radical prostatectomy as in stage 1, arm I.

Patients are followed at 1, 3, and 12 months.

PROJECTED ACCRUAL: A total of 20-80 patients (20 for stage 1 [10 per treatment arm] and 60 for stage 2) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Organ-confined disease
  * cT1, cT2, or cT3 tumors

    * Patients with cT1 tumors are eligible if ≥ 1 core biopsies have ≥ 50% of the tumor OR if 50% of the cores examined contain the tumor
  * No small cell carcinoma of the prostate
* Scheduled for radical prostatectomy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,500/mm^3

Hepatic

* ALT and AST ≤ 4 times normal
* Bilirubin ≤ 2 mg/dL

Renal

* Creatinine ≤ 2 times upper limit of normal
* Calcium ≤ 10.5 mg/dL
* No detectable renal stones by CT scan or ultrasound

Other

* No history of diabetes mellitus requiring pharmacotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* More than 5 years since prior antiestrogens, antiandrogens, luteinizing hormone-releasing hormone agonists, estrogen, or progestational agents

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* No prior nephrectomy
* No prior prostatic surgery
* No prior cryotherapy or transurethral resection of the prostate

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-09; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald L. Trump, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Patients receive oral dexamethasone once daily on days 1-4 and oral calcitriol once daily on days 2-4 weekly for 4 weeks before surgery.
  calcitriol: Given orally
  dexamethasone: Given orally
- Arm 2: No study drugs before surgery.
  clinical observation: No intervention before surgery
- Arm 3: Patients receive oral dexamethasone once daily on days 1-4.
  dexamethasone: Given orally
- Arm 4: Patients receive oral calcitriol once daily on days 2-4.
  calcitriol: Given orally
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 10 | 7 | 4 | 4
Completed | 9 | 7 | 4 | 4
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 10 | 7 | 4 | 4 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (7.8) | 56.3 (4.7) | 54.5 (8.3) | 50.2 (2.7) | 55.7 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 10 | 7 | 4 | 4 | 25

OUTCOME MEASURES:

1. Primary Outcome: Effect of Preoperative High-dose Calcitriol and Dexamethasone on Prostatic Tumor Vessel Density Measured at 1, 2, 3, and 12 Months Post Prostatectomy
Time Frame: Up to 30 days of the last administration of study procedure
Population: Study was activated in 9/2002 which was prior to Roswell Park Cancer Institute (RPCI) putting a system in place to centralize data entry and data management. Data entry of the outcomes was done by PI's staff and has since been lost. All attempts to retrieve the data have failed.
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Effect of Preoperative High-dose Calcitriol and Dexamethasone on Extent of Prostatic Intraepithelial Neoplasia (PIN) at 1, 2, 3, and 12 Months Post Prostatectomy
Time Frame: Up to 30 days of the last administration of study procedure
Population: as for outcome 1
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Determine the Effect of This Regimen on the Expression of Apoptosis Markers
Description: Determine the effect of this regimen on the expression of apoptosis markers, p21, p27, prostate-specific antigen (PSA), prostate-specific membrane antigen, and VDR expression in tumor-associated vascular endothelial cells and endothelium derived from normal-appearing prostate and tumor in these patients.
Time Frame: Up to 30 days of the last administration of study procedure
Population: as for outcome 1
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Determine the Acute Effects of This Regimen on Serum PSA in These Patients.
Time Frame: Up to 30 days of the last administration of study procedure
Population: as for outcome 1
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Adverse Events, Graded According to NCI CTCAE v2.0
Description: Number of Participants with Adverse Events, Graded According to NCI CTCAE v2.0
Time Frame: Up to 30 days of the last administration of study procedure
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 10 | 7 | 4 | 4
Participants
  Grade 1 | 1 | 2 | 2 | 2
  Grade 2 | 3 | 1 | 1 | 0
  Grade 3 | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/7 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 5/10 | 4/7 | 3/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=10) | Arm 2 (N=7) | Arm 3 (N=4) | Arm 4 (N=4)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=10) | Arm 2 (N=7) | Arm 3 (N=4) | Arm 4 (N=4)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was activated prior to Roswell Park Cancer Institute (RPCI) putting a system in place to centralize data entry and data management. Data entry was done by PI's staff. PI left institute and left incomplete data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes